CLINICAL TRIAL: NCT03079180
Title: Effect of Different Strength Training Intensities on Achilles and Patellar Tendon Adaptations With Aging
Brief Title: Tendon Adaptations to Training - Effect of Ageing
Acronym: TAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Université de Technologie de Compiegne (Other)
Collaborators: Centre Hospitalier Compiègne-Noyon (Unknown); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jean-Francois GROSSET, Associate Professor (PhD), Université de Technologie de Compiegne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016-A00534-47
Record Dates: First submitted 2017-02-09; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Aging; Exercise Training; Connective Tissue; Skeletal Muscle
Keywords: Tendon; Ageing; Training; Achilles tendon; Patella tendon; Skeletal muscle; Adaptation; Triceps Surae; Quadriceps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aged & strength training at 80% 1RM (Experimental): Subjects: 20 subjects aged between 65 and 85 years
  Training programs:
  Frequency: 3 training sessions per week. Duration: 12 weeks. Intensity: 80% of one repetition maximum (1RM). The 1RM of the participants in each of the 3 exercises performed in the training program will be reviewed every 2 weeks during training. If 1RM increase, the training load will be adjusted accordingly.
  Training exercises: A Warm-up will first be performed on a cycle ergometer during 10min. The training intervention will then consist in performing two sets on each one of the two exercises used for Patellar tendon stress: leg extension and leg press. To stress Achilles tendon, the subjects will perform four (4) sets using a calf raise machine. The subjects will perform 4 to 8 repetitions at 80% 1RM.
  All training sessions will take place under appropriate supervision in UTC for the duration of the interventions according to the study design.
  Interventions: Other: Strength training at 80% 1RM
- Aged & strength training at 55% 1RM (Experimental): Subjects: 20 subjects aged between 65 and 85 years
  The training program and training exercises in this group are the same as for the Aged & strength training at 80% 1RM arm except for the two following parameters.
  Training intensity: Intensity of exercises will be 55% of one repetition maximum (1RM).
  The subjects will perform 6 to 12 repetitions at 55% 1RM.
  The two training programs (55% or 80% of 1RM) are designed to be equal in volume (resistance x repetitions x sets).
  Interventions: Other: Strength training at 55% 1RM
- Young & strength training at 55% 1RM (Experimental): Subjects: 20 subjects aged between 18 and 30 years
  The training program and training exercises in this group are the same as for the Aged & strength training at 55% 1RM arm
  Interventions: Other: Strength training at 55% 1RM

INTERVENTIONS:
Other: Strength training at 80% 1RM — Detailed in Arms section's
  Arms: Aged & strength training at 80% 1RM
Other: Strength training at 55% 1RM — Detailed in Arms section's
  Arms: Aged & strength training at 55% 1RM; Young & strength training at 55% 1RM

SUMMARY:
Tendons are essential structures for transmitting muscle forces to skeletal structures. A stiffer tendon will transmit muscle force faster, and then allow faster movement. Moreover, tendons are a living tissue and respond to mechanical forces by changing their metabolism as well as their structural and mechanical properties. The aim of the present study is to answer essential questions remaining unanswered that are necessary in order to optimize physical activity with ageing in humans, and thus improve quality of life in elderly. The main questions are: What is the minimal training intensity leading to tendon adaptations? What is the time-course of tendon adaptations? Does the same loading protocol lead to similar tendon adaptations for different tendons (Achilles vs Patellar) and does the same training program lead to identical tendon adaptations with age (25yrs vs 75yrs)? To answer these questions, tendon architecture and mechanical properties will be investigated in humans of different age and applying different training intensities. The kinematic of the tendon adaptations due to these different training characteristics will also be investigated. The training protocol will be applied on plantar flexors and knee extensors. MRI and ultrasound techniques as well as the use of ankle and knee ergometers will allow the quantification of possible modifications in tendon architecture and mechanical properties (tendon stiffness and Young's Modulus). This will be assessed in vivo, using ultrasound images to assess tendon displacement during an incremental maximal contraction.

DETAILED DESCRIPTION:
Given the aging population demographics, and the barriers that exist in this population in terms of exercise participation, determining the level of exercise intensity required and the time-course to induce tendon adaptations is of paramount importance in this population. Therefore the purpose of this study is to:

1. determine whether a low intensity exercise training program (resistance 55% 1RM) affects tendon architecture and mechanical properties with aging,
2. compare these effects to those of a higher intensity exercise training protocol (resistance 80% 1RM) with a match training work with regards to the low intensity exercise training group,
3. evaluate the time course of tendon adaptations (architecture and mechanical properties) for the two training conditions with aging,
4. compare the effect of an identical training protocol applied on two different muscle groups (triceps surae vs quadriceps muscles) on Patellar and Achilles tendon adaptations.

Every subject recruited (Two groups composed of males aged between 65 and 85 years, and one group of young subjects (between 18 and 30 years)) will be asked to take part in a training program applied on the calf and quadriceps muscle groups on both legs. All subjects will be assessed 4 weeks before starting the intervention program (T-4w), at time zero (T0) and every four weeks during 12 weeks (T4w, and T8w). The investigation 4 weeks before starting the training program will allow using each subject as its own control. The intervention will involve a maximum of forty five (45) minutes training sessions 3 times per week. Subjects will be subjected to the same battery of baseline assessments (T-4w, and T0), during the training procedure (T4w, and T8w), and following the 12-weeks intervention period (T12w).

The effect of aging and different loading interventions on Achilles and Patellar tendon will be investigated for the following parameters:

* Tendon mechanical properties (stiffness and Young's Modulus) using US technique to assess Achilles and Patellar tendon displacement during an incremental maximal contraction.
* Tendon architecture using MRI technique to assess Achilles and Patellar tendon cross-sectional area, tendon length and moment arm.
* Maximal voluntary contraction (MVC)
* Muscle architecture using MRI technique.

Thus all these data will allow defining an optimal training intensity for physical activity of elderly persons.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age between 18 and 30 years for the young group and between 65 and 85 years for aged group
* Physical and mental health, as assessed by clinical investigation
* Written informed consent
* Willingness to co-operate
* Non-smoker
* Not addicted to alcohol or drugs
* Habitual sedentary/low physical activity levels

Exclusion Criteria:

* BMI <20 or >28
* Height <155cm, >195cm
* Chronic disease with regular clinical treatment
* Regular drug intake
* Any metabolic or hormonal disorder
* Psychiatric conditions
* Any blood clotting disorder
* Any muscle or bone disease
* Metal implants
* Any inflammatory disease
* Metabolic or hormonal disorder
* Participation in sports at competitive rather than at a recreational level
* Fractures during the past 6 months
* Epilepsy
* Back pain
* Lower extremity trauma during the past 6 months, or currently experiencing related symptoms, or receiving treatment
* Any other condition or history that the investigator considers might increase the risk to the individual or interfere with the evaluation of data

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-07-28 (Estimated); Study Completion 2017-07-28 (Estimated)

PRIMARY OUTCOMES:
Time-course change of tendon size | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Tendon size (tendon length and cross sectional area (CSA)) will be assessed using MRI.
Time-course change of tendon mechanics (Elastic modulus of the tendon) | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Tendon stiffness will be evaluated during voluntary plantar flexion contraction where force and elongation is measured using a force transducer and ultrasound, respectively. Tendon size will be assessed using MRI. Elastic modulus will be calculated based on stiffness and size of tendon.

SECONDARY OUTCOMES:
Time-course change of plantar flexion muscle strength | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Plantar flexion muscle strength will be assessed using a specifically designed ankle ergometer under isometric contraction.
Time-course change of calf muscle size | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Calf muscle size (i.e. cross sectional area and volume) will be assessed using MRI.
Time-course change of quadriceps muscle strength | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Quadriceps muscle strength will be assessed using a specifically designed knee ergometer under isometric contraction.
Time-course change of quadriceps muscle size | T-4weeks (4 weeks before starting intervention), T0 (before starting intervention), T+4weeks (after 4 weeks of intervention), T+8weeks (after 8 weeks of intervention), T+12weeks (at the end of the 12 weeks of intervention)
  Quadriceps muscle size (i.e. cross sectional area and volume) will be assessed using MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Franck Mabesoone, MD, Principal Investigator — Centre Hospitalier Compiegne-Noyon
Locations (1):
- Universite de Technologie de Compiegne, Compiègne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Letocart AJ, Mabesoone F, Charleux F, Couppe C, Svensson RB, Marin F, Magnusson SP, Grosset JF. Muscles adaptation to aging and training: architectural changes - a randomised trial. BMC Geriatr. 2021 Jan 13;21(1):48. doi: 10.1186/s12877-020-02000-0. PMID 33441116